CLINICAL TRIAL: NCT01742247
Title: Phase 4 Study of Assessment of Needs of Moisturizers After Various Laser Treatment
Brief Title: Assessment of Needs of Moisturizers After Various Laser Treatments
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PNUHDM-laser and moisturizers
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Dermatologic Disorders; Injury Due to Laser
Keywords: Moisturizer, laser
MeSH Terms: conditions — Skin Diseases | interventions — physiogel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physiogel, Laser therapy, Moisturizer (Experimental): Experimental: Physiogel treated & Non-treated
  1 Palmitoylethanolamide, Physiogel 3 times a day for 2 weeks
  Interventions: Other: Physiogel; Other: Moisturizer

INTERVENTIONS:
Other: Physiogel — Application of moisturizer on laser-treated area
  Other Names: Other moisturizer: Palmitoylethanolamide; Other Names:Physiogel
Other: Moisturizer — Application of moisturizer on laser-treated area
  Other Names: Other moisturizer: Palmitoylethanolamide; Other Names:Physiogel

SUMMARY:
Assessment of needs of moisturizers after various laser treatments

DETAILED DESCRIPTION:
The investigators would like to assess of needs of moisturizers after various laser treatment

: by investigating the changes in the skin barrier function after fractional carbon dioxide laser and fractional Er:Glass laser in mice and human skin

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age without any dermatologic diseases

Exclusion Criteria:

* Taking other known dermatologic disease
* Others who are shown pigmented lesion on treated-area
* Who have allergy or history of hypersensitivity reaction to moisturizers
* Who have other definitive cutaneous findings

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-09; Primary Completion 2015-04 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Clinical assessment of erythema, transepidermal water loss | 2weeks
  The clinical assessment of erythema, pigmentation, transepidermal water loss will be evaluated by using apparatus.

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Soo Kim, Ph.D., Study Chair — Pusna National University Hospital
Locations (1):
- Department of dermatology, Pusan National University Hospital, Busan, Busan, South Korea